CLINICAL TRIAL: NCT01668563
Title: International Subarachnoid Aneurysm Trial II Comparing Clinical Outcomes of Surgical Clipping and Endovascular Coiling for Ruptured Intracranial Aneurysms Not Included in the Original ISAT Study.
Brief Title: International Subarachnoid Aneurysm Trial II
Acronym: ISATII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE 12.136
Record Dates: First submitted 2012-08-15; First posted 2012-08-20 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Intracranial Hemorrhage Ruptured Aneurysm
Keywords: Aneurysm; Intracranial Aneurysm; Vascular Diseases; Cardiovascular Diseases; Intracranial Arterial Diseases; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases
MeSH Terms: conditions — Aneurysm; Intracranial Aneurysm; Vascular Diseases; Cardiovascular Diseases; Intracranial Arterial Diseases; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endovascular management (Active Comparator): Endovascular treatment will be performed as soon as possible following randomization, according to standards of practice, and under general anesthesia. Details regarding type of coils, use of adjunctive techniques such as balloon-remodeling, stents or flow-diverters, as well as post-treatment medical management issues, will be left up to the physician performing the endovascular treatment.
  Interventions: Procedure: Endovascular management
- Surgical management (Active Comparator): Surgical clipping will be performed as soon as possible following randomization, according to standards of practice, and under general anesthesia. Aneurysms thought by the treating physicians to require deliberate permanent proximal vessel occlusion, construction of a surgical bypass, or other flow-redirecting treatments that do not directly clip the aneurysm will not be excluded; these non-ISAT aneurysms are expected to be more difficult lesions to manage surgically as well as endovascularly.
  Interventions: Procedure: surgical management

INTERVENTIONS:
Procedure: surgical management — Surgical clipping will be performed as soon as possible following randomization, according to standards of practice, and under general anesthesia. Aneurysms thought by the treating physicians to require deliberate permanent proximal vessel occlusion, construction of a surgical bypass, or other flow-redirecting treatments that do not directly clip the aneurysm will not be excluded; these non-ISAT aneurysms are expected to be more difficult lesions to manage surgically as well as endovascularly.
  Arms: Surgical management
Procedure: Endovascular management — Endovascular treatment will also be performed as soon as possible following randomization,according to standards of practice, and under general anesthesia. Details regarding type of coils, use of adjunctive techniques such as balloon-remodeling, stents or flow-diverters, as well as post-treatment medical management issues, will be left up to the physician performing the endovascular treatment.
  Arms: Endovascular management

SUMMARY:
The purpose of this study is to compare the clinical outcome of surgical clipping and endovascular coiling for ruptured intracranial aneurysms not included in the original ISAT Study.

DETAILED DESCRIPTION:
The International Subarachnoid Aneurysm Trial (ISAT) was a turning point in modern neurosurgical history (1). The trial showed that for 2143 subarachnoid hemorrhage (SAH)patients eligible for both surgery and endovascular coiling, randomized allocation to coiling was associated with better one year clinical outcomes, defined as survival without dependency (absolute risk reduction (ARR) of 7.4% (95%CI; 3.6 - 11.2, p=0.0001). Because ISAT was a positive pragmatic trial, the interpretation of the trial results was that coiling should be adopted as the first-line treatment for ruptured lesions, for patients with the types of aneurysms included in ISAT, of which the great majority were small (≥10 mm) anterior circulation aneurysms.

Although ISAT was well-designed, conducted, and reported, trial results were not always properly interpreted, and endovascular coiling was perhaps inappropriately extrapolated beyond what ISAT demonstrated. Endovascular treatment for ruptured aneurysms has now become first-line treatment in many centers (2), which may be appropriate for small, anterior circulation lesions, but there is no evidence to support this practice for the wide spectrum of non-ISAT patients and aneurysms. A recent pre-randomized study of coiling as first-intention (3)showed better results for those ruptured aneurysms felt to be readily coilable; however, the optimal management of more difficult-to-coil ruptured aneurysms remains unclear.

Further compounding the problem are the concerns that aneurysm coiling may not be as durable in the long-term as surgical clipping, leading many neurosurgeons to continue to clip most ruptured aneurysms in spite of ISAT results.

Proponents of endovascular treatment sometimes justify this extrapolation of ISAT results on the basis of improved catheter and coil technology, although this has never been demonstrated. However, the addition of stents and flow-diverters, which were not tested in ISAT, may increase endovascular treatment risks, especially when combined with dual anti-platelet agents. The introduction of these devices allowed for the expansion of indications of EVT to include wide-necked aneurysms, lesions which would not have been included in ISAT. The wider spectrum of patients and aneurysms now considered for EVT may not all experience the same degree of benefit as seen in the original ISAT trial (4). Considering the relatively small ARR of 7.4% favouring coiling, when the additional risks due to stents are included, the balance may have tipped to favour surgical clipping.

These new questions deserve formal study in the context of a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* At least one documented, intradural, intracranial aneurysm, ruptured within last 30 days
* SAH WFNS grade 4 or less
* The patient and aneurysm are considered appropriate for either surgical or endovascular treatment by the treating team

Exclusion Criteria:

* Patients with absolute contraindications administration of contrast material (any type)
* Patients with AVM-associated aneurysms
* Aneurysm located at basilar apex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1724 (Estimated)
Dates: Start 2012-11-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
poor clinical outcome(mRS>2) | 12 months
  Number of patients experiencing a poor clinical outcome at one year post-treatment, defined as a modified Rankin Scale (mRS) score of >2.

SECONDARY OUTCOMES:
Occurrence of an intracranial hemorrhage following treatment | one year
  An intracranial hemorrhage will be judged from cross-sectional imaging (CT or MRI), from a positive lumbar puncture in the setting of an acute headache, or following sudden death preceded by an acute headache.
Failure of aneurysm occlusion using the intended treatment modality | within 48 hours after attempted treatment
  In situations where treatment is initiated but terminated without a proper test of that treatment modality, such as in the event of anaesthetic difficulty requiring the intended treatment to be delayed, will not count as a failure. However, patients left with clinically concerning aneurysm residuals (in the opinion of the treating physician) after the treatment attempt will count as a failure of the initial treatment.
Overall mortality and morbidity | one year and five years
  Mortality and morbidity from all causes will be recorded, along with cause of death, at one and five years.
Occurence of a "major" (saccular) aneurysm recurrence | 12 months (+/- 2 months)
  Determined using non-invasive angiography (CTA or MRA)as part of normal follow-up after aneurysm treatment. Although DSA, CTA and MRA are known to have different sensitivities in detecting aneurysm remnants,these modalities are equally well-suited to the discovery of a concerning, saccular aneurysm residual or remnant.
Peri-treatment hospitalization lasting more than 20 days and/or discharge to a location other than home | within a month or at discharge if earlier
  Will be recorded by the local treating physician upon discharge.
Occurence of aneurysm re-rupture following randomization but before treatment initiation | Within a few hours (while awaiting treatment)
  Repeat intracranial hemorrhage will be judged from cross-sectional imaging (CT scan), after worsening of headache, or following a new-onset neurological deficit or sudden death while awaiting treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Darsaut, MD, Principal Investigator — University of Alberta; Max Findlay, MD, Principal Investigator — University of Alberta
Locations (6):
- Montefiore Medical Center, The Bronx, New York, United States
- Canada (3):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Centre Hospitalier de l'Université de Montréal - Hôpital Notre Dame, Montreal, Quebec
- Spain (2):
  - Vall d'Hebron Hospital, Barcelona
  - University of Valladolid, Valladolid

REFERENCES:
- [Background] Molyneux A, Kerr R, Stratton I, Sandercock P, Clarke M, Shrimpton J, Holman R; International Subarachnoid Aneurysm Trial (ISAT) Collaborative Group. International Subarachnoid Aneurysm Trial (ISAT) of neurosurgical clipping versus endovascular coiling in 2143 patients with ruptured intracranial aneurysms: a randomised trial. Lancet. 2002 Oct 26;360(9342):1267-74. doi: 10.1016/s0140-6736(02)11314-6. PMID 12414200
- [Background] Gnanalingham KK, Apostolopoulos V, Barazi S, O'Neill K. The impact of the international subarachnoid aneurysm trial (ISAT) on the management of aneurysmal subarachnoid haemorrhage in a neurosurgical unit in the UK. Clin Neurol Neurosurg. 2006 Feb;108(2):117-23. doi: 10.1016/j.clineuro.2005.11.001. Epub 2005 Dec 20. PMID 16364540
- [Background] McDougall CG, Spetzler RF, Zabramski JM, Partovi S, Hills NK, Nakaji P, Albuquerque FC. The Barrow Ruptured Aneurysm Trial. J Neurosurg. 2012 Jan;116(1):135-44. doi: 10.3171/2011.8.JNS101767. Epub 2011 Nov 4. PMID 22054213
- [Background] Raymond J, Kotowski M, Darsaut TE, Molyneux AJ, Kerr RS. Ruptured aneurysms and the International Subarachnoid Aneurysm Trial (ISAT): What is known and what remains to be questioned. Neurochirurgie. 2012 Apr-Jun;58(2-3):103-14. doi: 10.1016/j.neuchi.2012.02.020. Epub 2012 Apr 4. English, French. PMID 22481029
- [Derived] Darsaut TE, Jack AS, Kerr RS, Raymond J. International Subarachnoid Aneurysm Trial - ISAT part II: study protocol for a randomized controlled trial. Trials. 2013 May 29;14:156. doi: 10.1186/1745-6215-14-156. PMID 23714335